CLINICAL TRIAL: NCT04193800
Title: The Effect of a Specialist Paramedic Primary Care Rotation on Appropriate Non-conveyance Decision: a Controlled Interrupted Time Series Analysis
Brief Title: Specialist Paramedic Rotations And Their Impact on Non-conveyancE Decisions
Acronym: SPRAINED
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yorkshire Ambulance Service NHS Trust (Other Government)
Collaborators: Applied Research Collaboration for Yorkshire and Humber (Unknown)
Responsible Party: Sponsor
Other Study IDs: YASRD128
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Safe Paramedic Non-conveyance
MeSH Terms: interventions — Rotation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rotational paramedic pilot group
  Interventions: Other: 10-week rotation in primary care setting
- Paramedic control group

INTERVENTIONS:
Other: 10-week rotation in primary care setting — Ten paramedics underwent a 10 week rotation into a GP practice in the Leeds area of South Yorkshire, England.
  Groups: Rotational paramedic pilot group

SUMMARY:
The National Health Service (NHS) in the United Kingdom is facing a 5% increase in demand every year for urgent and emergency care services, and there is evidence that patients are being taken to hospitals by ambulance services when they do not need to go. This is a problem because emergency departments are becoming more crowded, which can lead to poorer quality care. Also, less ambulances are available to respond to emergencies, because they are queueing at hospital for a long time.

To improve the care Yorkshire Ambulance Service provide to their patients, some paramedics have received additional training. These advanced paramedics have been very successful at treating patients in their own home safely. However, their training is long and expensive, so another role, the specialist paramedic role has been introduced. Their training does not take as long and is cheaper to provide. However, the specialist paramedics do not appear to keep patients safely at home more often than regular paramedics. Recently, the specialist paramedics have taken part in a national paramedic programme, where they are given the chance to work in GP surgeries and emergency call centres.

This study aims to see if specialist paramedics who have worked in a GP surgery for 10 weeks, can keep patients at home safely, and without costing too much, more often than regular paramedics.

DETAILED DESCRIPTION:
The National Health Service (NHS) in the United Kingdom is facing a 5% year-on-year increase in demand for urgent and emergency care services. In 2018/19, ambulance services in England provided a face-to-face assessment to nearly 7.9 million incidents, of which 7.6 million were conveyed to hospital. This conveyance rate of around 69% is occurring despite an increase in urgent cases and is placing increasing demands on already crowded emergency departments (EDs), leading to decreased availability of ambulances as turnaround times at hospitals increase. ED overcrowding is a significant issue for patients, resulting in poorer quality of care, increased healthcare costs and potentially, increased mortality.

Yorkshire Ambulance Service have been early adopters of initiatives to address inappropriate conveyance, and have had paramedics working in the role of Emergency Care Practitioners (ECP), since 2004. ECPs consistently have non-conveyance rates double that of other paramedics in the Trust. More recently, the specialist paramedic (SP) role has been introduced, although the educational programme is less substantial than that of the ECPs, and non-conveyance rates have been no different to other paramedics within the Trust.

In 2018, Health Education England funded a pilot scheme to rotate paramedics into a range of healthcare settings, with the aim of improving patient care and relieving pressures on primary care, ambulance services and other parts of the NHS in a sustainable way. This pilot also presents an opportunity to develop SPs and potentially, improve their rates of appropriate non-conveyance which may deliver patient and cost-benefits of the role as originally anticipated.

This study aims to evaluate whether the paramedics who have rotated into primary care, are appropriately and cost-effectively increasing the level and trend of non-conveyance decisions compared to a matched control population of YAS paramedics.

This study will use a dataset comprised of non-identifiable, routinely collected, ambulance service data to undertake a controlled interrupted time series analysis. This is one of the strongest quasi-experimental designs to detect change in the level and trend of paramedic appropriate non-conveyance decisions. The cost-effectiveness analysis will examine the cost per appropriate non-conveyance achieved for patients receiving care from paramedics who have completed a 10-week rotation in a GP surgery compared with those receiving care from paramedics who did not take part in the primary care rotational pilot.

ELIGIBILITY:
Inclusion Criteria:

* Incident date 12 months before or after the 10 week rotational pilot period
* Adult patient receiving a face-to-face assessment by a paramedic taking part in the primary care rotation pilot, or
* Matched adult patient who receive a face-to-face assessment by a paramedic not taking part in the rotation pilot
* Has a completed paper or electronic patient care record.

Exclusion Criteria:

* Patient under the age of 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All face-to-face patient care episodes that were attended by one of the 10 rotational paramedics between the 1st June, 2017 to 31st December, 2019 and an additional cohort of patients who have receive a face-to-face assessment by paramedics who have not taken part in the GP rotation.
Sampling Method: Non-Probability Sample
Enrollment: 33600 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-01-02 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in proportion and trend of safe non-conveyance | 12 months
  Change in proportion of appropriate non-conveyance decision by paramedics immediately following a 10-week rotation in a GP surgery, and the trend in non-conveyance decision in the 12-month period following the rotation

CONTACTS AND LOCATIONS:
Locations (1):
- Yorkshire Ambulance Service NHS Trust, Wakefield, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to make this dataset available to other researchers.